CLINICAL TRIAL: NCT04607070
Title: Ischemic Strokes While on NOAC - How Compliance Matters
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Specialist resident, Chinese University of Hong Kong
Other Study IDs: Crec 2020.427
Record Dates: First submitted 2020-10-23; First posted 2020-10-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Ischemic; Stroke, Acute; Stroke Syndrome; Stroke, Cardiovascular; Atherosclerosis; Ischemic Stroke
Keywords: stroke, NOAC
MeSH Terms: conditions — Ischemic Stroke; Stroke; Myocardial Infarction; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patient: This is a registry-based study that will involve consecutive adult patients with known AF who developed ischaemic stroke or TIA in years 2010, 2012, 2014, 2016 and 2018.

SUMMARY:
This study is aimed to depict the epidemiological trend, aetiologies, clinical characteristics, treatment options of IS-NOAC in face of the rapidly increasing NOAC usage. Knowledge on this ischaemic stroke entity will define clinical characteristics, identify preventable causes and inform resource allocation on the evaluation modalities, reperfusion strategies and forecast future burden of IS-NOAC.

DETAILED DESCRIPTION:
Data will be retrieved from the stroke registry of Prince of Wales Hospital which recorded all in- and out-patients with stroke or transient ischaemic attack (TIA). All consecutive adult patients with known AF who developed ischaemic stroke or TIA in 2010, 2012, 2014, 2016 and 2018 (i.e. 5 full yearly time-points) and categorize the patients according to their anticoagulation status (elaborated below) with the inclusion and exclusion criteria stated will be recruited.

All demographic data, blood results, imaging and assessment data will be retrieved from electronic patient record (CMS system) and stroke registry. All-cause mortality at 1 year will be verified via CMS system too.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were ethnic Chinese
2. Patients with known AF
3. Patient who suffered from ischaemic stroke

Exclusion Criteria:

1. Patient who are non-ethnic Chinese
2. Patient who suffered from haemorrhagic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known AF who developed ischaemic stroke or TIA and admitted in the Prince of Wales Hospital in years 2010, 2012, 2014, 2016 and 2018 will be recruited into this study
Sampling Method: Non-Probability Sample
Enrollment: 870 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Compliance affects the outcomes of ischemic stroke during NOAC usage. | 30 Sept 2021
  To depict epidemiological trend and aetiologies on different dosage of NOAC in stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Ming Bonaventure IP, MBChB, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No